CLINICAL TRIAL: NCT06982573
Title: The Effect of Magnetic Stimulation on Low Back Pain Relief and Muscle Mass Maintenance in Patients With End-Stage Renal Disease (ESRD)
Brief Title: The Effect of Magnetic Stimulation on Low Back Pain Relief and Muscle Mass Maintenance in Patients With ESRD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bundang CHA Hospital (Other)
Responsible Party: Principal Investigator, MinYoung Kim, MD, PhD, Principle investigator, Bundang CHA Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2025-01-031
Record Dates: First submitted 2025-05-11; First posted 2025-05-21 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: End-Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- End-Stage Renal Disease patients (Experimental)
  Interventions: Device: Effects of applying magnetic stimulation

INTERVENTIONS:
Device: Effects of applying magnetic stimulation — The Effect of Magnetic Stimulation on Low Back Pain Relief and Muscle Mass Maintenance in Patients with End-Stage Renal Disease (ESRD)

SUMMARY:
To determine the effectiveness of magnetic stimulation application on alleviating back pain and maintaining muscle mass in patients with end-stage renal disease.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 19 years or older
2. Patients diagnosed with end-stage renal failure and receiving dialysis treatment more than three times a week
3. Back pain intensity of 4 points or higher on the visual analogue scale (VAS)
4. Those with cognitive function that can clearly indicate NRS with a score of 23 points or higher, the criterion for determining cognitive impairment on the Mini Mental State Examination (MMSE) [14]
5. Those who voluntarily decided to participate in this clinical trial after receiving a detailed explanation and fully understanding it and gave written consent to comply with the precautions

Exclusion Criteria:

1. If the pain is due to trauma
2. If it is difficult to participate in the study due to serious mental illness (e.g. schizophrenia, bipolar disorder, etc.) or psychological instability.
3. Patients with severe neurological illness (e.g. stroke, severe dementia, etc.).
4. Those with poor general condition due to unstable cardiovascular, digestive, respiratory, or endocrine systems, or severe internal medical illness such as systemic infection
5. Patients participating in other therapeutic clinical trials or those who have participated in other therapeutic clinical trials within the past 30 days (observational studies are not relevant)
6. If there are contraindications to magnetic stimulation

   * Patients with implanted medical devices (e.g. pacemakers)
   * Metal objects are inserted into the skull
   * A wound on the skin at the attachment site
   * History of epilepsy
   * Cervical pain or musculoskeletal disease
   * Pregnant and lactating women

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2026-02-19 (Estimated); Study Completion 2026-02-19 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Sclae (VAS) | 7 days before intervention/1 day after intervention/1 month after intervention
  An assessment in which the subject quantifies the level of pain numerically from 0 to 10. The higher the number, the more intense the pain.

SECONDARY OUTCOMES:
Short Physical Performance Battery (SPPB) | 7 days before intervention/1 day after intervention/1 month after intervention
  Measures balance, lower extremity strength, and functional ability on a scale of 0 to 16. Higher scores indicate better function.
The World Health Organization (WHOQOL-BREF) | 7 days before intervention/1 day after intervention/1 month after intervention
  The WHOQOL-BREF consists of 26 items, with scores ranging from 1 to 5. A higher score indicates a higher quality of life.
3D Motion Capture | 7 days before intervention/1 day after intervention/1 month after intervention
  Collecting human body movement data using a 3D infrared camera and ground reaction force device
Dual Energy X-ray Absorptionmetry (DEXA) | 7 days before intervention/1 day after intervention/1 month after intervention
  A test that measures muscle mass by utilizing the energy absorption properties of high-energy and low-energy X-rays.

CONTACTS AND LOCATIONS:
Overall Officials: Kim Minyoung, M.D., Ph.D, Principal Investigator — Bundang CHA Hospital
Locations (1):
- CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No